CLINICAL TRIAL: NCT03954613
Title: Evaluation of the Contribution of Regular Cognitive Exercises to Treatment in Patients With Alzheimer's Disease Receiving Donepezil, Memantine or Donepezil/Memantine Combination Therapy: Open-Labeled, Randomized, Phase IV, Superiority Study
Brief Title: Evaluation of the Contribution of Regular Cognitive Exercises to Treatment in Patients With Alzheimer's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU-05.18
Record Dates: First submitted 2019-04-09; First posted 2019-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Alzheimer Disease; Cognitive Change
Keywords: Alzheimer Disease; Cognitive Exercises; Internet; Donepezil; Memantin; Combination
MeSH Terms: conditions — Alzheimer Disease | interventions — Namzaric

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A (Experimental): Donepezil/Memantin Combination
  Interventions: Combination Product: Ebicomb
- Group B (Experimental): Donepezil/Memantin Combination + Cognitive Exercises (BEYNEX Software)
  Interventions: Combination Product: Ebicomb
- Group C (Active Comparator): Donepezil Mono
  Interventions: Combination Product: Ebicomb
- Group D (Active Comparator): Donepezil Mono + Cognitive Exercises (BEYNEX Software)
  Interventions: Combination Product: Ebicomb
- Group E (Active Comparator): Memantine Mono
  Interventions: Combination Product: Ebicomb
- Group F (Active Comparator): Memantine Mono + Cognitive Exercises (BEYNEX Software)
  Interventions: Combination Product: Ebicomb

INTERVENTIONS:
Combination Product: Ebicomb — Combination product and combination product plus cognitive exercises will primarily be evaluated in this study
  Other Names: Donepezil-Memantine

SUMMARY:
In this study, it is aimed to compare the effects of cognitive exercises applied on long-term internet environment to the cognitive level of patients who received donepezil, memantine or donepezil / memantin combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 55-90 years old who were diagnosed with Alzheimer's Dementia and had no history of cerebrovascular disease during the last 6 months,
* Patients without other neurodegenerative diseases and secondary dementia diagnoses,
* Patients with MOCA score of between 13-18,
* Patients with at least primary school graduation,
* Patients who have had no CNS disease including trauma in the last year,
* Patients without a diagnosis of psychiatric disease,
* Patients with a tablet or PC with an internet connection,
* Patients agreeing to perform BEYNEX daily activity at least 5 times per week,
* Patients signing informed consent form.

Exclusion Criteria:

* Patients who have hypersensitivity to study working drugs,
* Psychotic patients,
* Disabled patients with orthopedic dominant extremity,
* Patients with ICU follow-up due to trauma in the last 6 months,
* Patients with severe visual impairment or eye surgery,
* Patients who refuse to sign the informed consent form.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in MOCA total score | 6-months
  MOCA: Montreal - Cognitive Assessment

SECONDARY OUTCOMES:
Change in GDS total score | 6-months
  GDS (The Geriatric Depression Scale)
Change in ADAS-Cog total score | 6-months
  ADAS-Cog: Alzheimer's Disease Assessment Scale- Cognitive Subscale
Change in CDR total score | 6-months
  CDR: The Clinical Dementia Rating
Change in B-ADL total score | 6-months
  B-ADL: The Bayer Activities of Daily Living Scale
Change in clock drawing test | 6-months
  The subject is asked to draw the face of a clock with all numbers and to set the hands for a specified time (hh:mm) and will be evaluated according to ability to draw.

CONTACTS AND LOCATIONS:
Overall Officials: Türker Şahiner, Prof Dr, Study Chair — Project Consultant
Locations (1):
- Maltepe University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided